CLINICAL TRIAL: NCT04005703
Title: Whole-body MRI for Initial Staging, Early Response Assessment and Restaging After Completion of Therapy in Pediatric Hodgkin's Lymphoma.
Brief Title: Whole-body MRI in Pediatric Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Stichting Kinderen Kankervrij (KiKa) (Unknown)
Responsible Party: Principal Investigator, R.A.J. Nievelstein, Principal Investigator, UMC Utrecht
Other Study IDs: KIKA project number 87
Record Dates: First submitted 2013-07-02; First posted 2019-07-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hodgkin's Lymphoma
Keywords: Malignant lymphoma; Hodgkin's disease; Imaging; Whole-Body MRI; PET/CT; Radiation
MeSH Terms: conditions — Hodgkin Disease; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Hodgkin's lymphoma: Children with newly diagnosed Hodgkin's lymphoma

SUMMARY:
Background:

The assessment of extent of disease (staging) and response to therapy (restaging) is performed with computed tomography (CT) scan, 18F-fluorodeoxyglucose positron emission tomography (FDG-PET scan) or integrated FDG-PET/CT. Whole-body MRI with diffusion weighted imaging (WB-MRI with DWIBS) is a radiation-free method which allows imaging of the body with excellent soft tissue contrast in a single examination and could be an attractive alternative to FDG-PET and CT for the staging and restaging of malignant lymphomas in children.

Aim of the study:

The aims of this study are to compare the diagnostic performance of whole-body MRI (including DWIBS) to FDG-PET/CT and/or CT for the initial staging, early response assessment and restaging after completion of therapy in children with Hodgkin's lymphoma.

Study design:

Patients eligible for enrollment in this multicenter, prospective, diagnostic cohort study are children aged 8-18 years, with histologically confirmed Hodgkin's lymphoma, who are treated according to the EuroNet-PHL-C1 protocol (or trial with similar imaging strategy) in one of the participating centers. Patients will undergo WB-MRI in addition to the protocolar imaging routinely done (FDG-PET(/CT) and CT scan) at 3 time-points: at initial staging, after 2 chemotherapy cycles and at end of treatment. The investigators expect to enrol 75 patients in a 3 year study period. Staging and restaging results of WB-MRI (according to the Ann Arbor and Cheson classification, respectively) will be compared to those of FDG-PET(/CT) and CT. Clinical and radiological follow-up after 6 months will be used to solve any disagreements between FDG-PET, CT and WB-MRI. Additionally, the investigators will collect 3 year follow-up clinical data and data on follow-up imaging from the hospital charts of the patients, to better assess the prognostic value of FDG-PET and WB-MRI.

DETAILED DESCRIPTION:
Background:

The malignant lymphomas, Hodgkin´s lymphoma (HL) and non-Hodgkin´s lymphoma (NHL), comprise approximately 10% of childhood cancers. The assessment of extent of disease (staging) and response to therapy (restaging) is performed with computed tomography (CT) scan, 18F-fluorodeoxyglucose positron emission tomography (FDG-PET scan) or integrated FDG-PET/CT. Staging and restaging are important for choice of treatment and for determining prognosis. Unfortunately, FDG-PET and CT are accompanied by a significant amount of radiation exposure which may induce second cancers. New magnetic resonance imaging (MRI) techniques offer an alternative way for staging and follow-up of cancers. Whole-body MRI with diffusion weighted imaging (WB-MRI with DWIBS) is a radiation-free method which allows imaging of the body with excellent soft tissue contrast in a single examination and could be an attractive alternative to FDG-PET and CT for the staging and restaging of malignant lymphomas in children.

Aim of the study:

The aims of this study are to compare the diagnostic performance of whole-body MRI (including DWIBS) to FDG-PET/CT and/or CT for the initial staging, early response assessment and restaging after completion of therapy in children with Hodgkin's lymphoma.

Study design:

Patients eligible for enrollment in this multicenter, prospective, diagnostic cohort study are children aged 8-18 years, with histologically confirmed Hodgkin's lymphoma, who are treated according to the SKION / EuroNet-PHL-C1 protocol (or trial with similar imaging strategy) in one of the participating centers. Patients will undergo WB-MRI in addition to the protocolar imaging routinely done (FDG-PET(/CT) and CT scan) at 3 time-points: at initial staging, after 2 chemotherapy cycles and at end of treatment. We expect to enrol 75 patients in a 3 year study period. Staging and restaging results of WB-MRI (according to the Ann Arbor and Cheson classification, respectively) will be compared to those of FDG-PET(/CT) and CT. All imaging modalities will be assessed by a radiologist and nuclear medicine physician in a blinded fashion, using standardized score forms. Findings of FDG-PET and CT together will serve as the reference standard. Clinical and radiological follow-up after 6 months will be used to solve any disagreements between FDG-PET, CT and WB-MRI. Additionally, at least 3 year follow-up clinical data and data on follow-up imaging will be collected from the hospital charts of the patients, to better assess the prognostic value of FDG-PET and WB-MRI.

Clinical/scientific relevance:

This study aims to assess the accuracy of WB-MRI compared to FDG-PET(/CT) and CT in staging and response assessment of Hodgkin lymphoma. The results of this study can contribute to the development of evidence based 'radiation reduced' imaging protocols in Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* age: 8-18 years
* histologically proven Hodgkin's lymphoma
* enrolled in the EuroNet-PHL-C1 trial (or trial with comparable imaging strategy)
* patients scheduled for a FDG-PET/CT and/or CT of the body for initial staging, early response assessment (after two cycles of chemotherapy) or restaging
* participant's parents (and participants >12 years of age) must willingly give written informed consent prior to each MRI
* whole-body MRI/DWIBS has to be performed within 15 days before or after FDG-PET/CT or CT and the initial staging MRI should be performed before therapy has been started

Exclusion Criteria:

* patients with a general contraindication for MRI (including cardiovascular pacemakers, claustrophobia)
* patients who have had a previous malignancy
* patients who are pregnant or nursing
* patients in whom therapy has already started after FDG-PET/CT and/or CT and before the initial WB-MRI/DWIBS could be performed
* apparent signs of resistance during MR examination

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients, aged 8-18 years, with newly diagnosed Hodgkin's lymphoma, who will undergo PET/CT for staging, early response assessment and restaging at completion of therapy (imaging standards according to the Euronet-PHL-C1 protocol).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Staging (Ann Arbor) | Day 1
  The primary outcome parameter will be the clinical stage according to WB-MRI (including DWIBS) and according to FDG-PET/CT. This clinical stage will be determined according to the Ann Arbor classification system for initial staging.
Early treatment response assessment (Cheson criteria) | 2 months
  The primary outcome parameter will be the clinical stage according to WB-MRI (including DWIBS) and according to FDG-PET/CT. This clinical stage will be determined according to the Cheson criteria for early response assessment.
Restaging at end of therapy (Cheson criteria) | 6 months
  The primary outcome parameter will be the clinical stage according to WB-MRI (including DWIBS) and according to FDG-PET/CT. This clinical stage will be determined according to the Cheson criteria for restaging.
Follow up for 3 years after end of treatment | 3 years
  The percentage of relapse of Hodgkin lymphoma in this study cohort will be assessed by a 3-year follow-up of clinical and imaging data, and the percentage of true- versus false-positives on WB-MRI at end of treatment compared to PET/CT using this follow-up.

SECONDARY OUTCOMES:
Image quality | Day 1, 2 months, 6 months
  The secondary outcome will be a (subjective) assessment of image quality and presence of artefacts, for both T1-weighted and T2-weighted MR images, MR-DWI as well as PET/CT.
Interobserver variability of WB-MRI for staging, early response assessment and restaging at end of therapy | Day 1, 2 months, 6 months
  The interobserver variability of WB-MRI (including DWIBS) for staging, early response assessment and restaging at end of therapy will be determined for two observers.

CONTACTS AND LOCATIONS:
Overall Officials: Rutger AJ Nievelstein, MD PhD, Principal Investigator — UMC Utrecht
Locations (8):
- LKH-Universitätsklinikum Graz, Graz, Austria
- Ospedale Giannina Gaslini, Genova, Italy
- Netherlands (5):
  - Academic Medical Center Amsterdam, Amsterdam
  - VU University Medical Center, Amsterdam
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- HUMI Vall d'Hebron, Barcelona, Spain